CLINICAL TRIAL: NCT01906684
Title: Comprehensive Analysis of Relapse in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanner Foundation for Multiple Sclerosis (Other)
Collaborators: Mallinckrodt (Industry); Auburn University MRI Research Center (Unknown); iReportoire Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFMS:QP1-2013
Record Dates: First submitted 2013-07-19; First posted 2013-07-24 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Sclerosis
Keywords: Acthar Gel; MS relapse; 7T MRI imaging; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acthar Gel (Experimental): Acthar Gel is supplied as 5 mL multi-dose vial (63004-8710-1) containing 80 USP Units per mL. H.P. Acthar Gel (repository corticotropin injection). Acthar Gel will be administered as a subcutaneous daily dose of 80 units for up to 2 weeks.
  Interventions: Drug: Acthar Gel

INTERVENTIONS:
Drug: Acthar Gel — Patients who present with MS relapse within 72 hours of onset will be recruited for study. Upon consent they will be administered Achtar Gel for 5-14 days as clinically appropriate.

SUMMARY:
This study will determine changes in: 1) the immune activity, characterized as the "immunorepertoire;" 2) 7 Tesla MRI brain images; 3) clinical outcomes; and 4) patient reported quality of life outcomes in subjects with relapsing-remitting multiple sclerosis who are treated with Acthar Gel.

DETAILED DESCRIPTION:
20 patients with documented Multiple Sclerosis, who have been diagnosed within 12 months of enrollment in the study and who are currently experiencing an MS relapse, defined as the following manifestation:

Acute onset or worsening of any of the manifestations of CNS relapses (excluding spinal cord) including:

* Brain stem syndrome
* Optic neuritis
* Cerebellar syndromes

If they choose to participate, subjects will be asked to:

Meet at the Clinic 4 times:

* Initial visit
* 5 days after baseline visit
* 14 days after baseline visit
* 30 days after baseline visit

Meet with neurologist for neurological exam that will include a:

* Review of neurological status
* Review of new and ongoing symptoms
* Review of symptom resolution
* Review of any side effects or adverse events
* Resolution of any patient questions and concerns
* Provide a 40cc whole blood sample

At each of the 4 visits

* Consent to Acthar Gel treatment for their relapse for 14 days (or as required for their relapse)
* Ss will agree to be trained in self-administration of Acthar
* First dose administered at Baseline visit
* Self-administered days 2-14 of participation
* Complete 4 psychometric instruments

At baseline and 30 day visit

* Cognitive assessment using the Brief International Cognitive Assessment for MS (Benedict 2012)
* Administered by Tanner Center Staff specially trained in this assessment
* Quality of Life assessments: self-administered
* MSQoL (Cella et al, 1006)
* Psychological Adjustment to Illness Survey (Rodrigue et al 2000)
* Coping Skills Inventory (Liveneh, 2003)
* Participate in a brief semi-structured interview, at Day 5 visit

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate in the study if:

They were diagnosed with Relapsing-Remitting Multiple Sclerosis within 1 year of their participation in the study Are established patients of the Tanner Center for MS Seek care for relapse within 72 hours of onset Are between the ages of 19 and 65 inclusively.

Relapse will be confirmed and defined as the acute worsening of function that lasts for at least 24 hours with any of the manifestations of Central Nervous System relapses (excluding spinal cord) including:

Brain stem syndrome Optic neuritis Cerebellar syndromes Hemi-motor/sensory events Males and Females are both eligible Patients of any race or ethnicity are eligible Are not pregnant (as confirmed by pregnancy test at the time of enrollment) or nursing Have no known contraindicating conditions (see exclusions)

Exclusion Criteria:

* Potential participants will be excluded if they do not meet the above criteria, and also if:

They are currently being treated for MS with the any of the following disease-modifying drugs: Tysabri, Gilenya, Aubagio, Tecfidera They have a history of experiencing significant adverse reactions to corticosteroids They are deemed by Dr Riser to be better served with an intervention other than Acthar Gel to treat their current MS relapse Are pregnant or nursing

Are known to have any of the contraindicating conditions:

Scleroderm Osteoporosis Systemic fungal infections Ocular herpes simplex Recent surgery History of or presence of peptic ulcer Congestive heart failure Uncontrolled hypertension Adreno-cortical insufficiency, hyper-function or sensitivity Sensitivity to proteins of porcine origin

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Changes in immunorepertoire, MRI imaging, clinical outcomes and patient reported quality of life | within 1 month post initiation of treatment with Acthar Gel
  This study will observe changes in the activity of b cells and t cells as evidenced in the patient's immunorepertoire, as well as changes in 7T MRI images, physician-documented clinical outcomes in patients receiving Acthar Gel for treatment of MS relapse at four time points: baseline, 5, 14 and 30 days post initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Emily S Riser, MD, Principal Investigator — Tanner Center for MS
Locations (1):
- Tanner Center for MS, Birmingham, Alabama, United States